CLINICAL TRIAL: NCT06643026
Title: Sensory Evaluation of Taste and Smell in Oncology
Acronym: SENSEO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0728
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Digestive Cancers
Keywords: digestive cancers; chemotherapy; food preference; sensory perceptions
MeSH Terms: conditions — Gastrointestinal Neoplasms; Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with digestive cancer traited by chemotherapy: Patients with malignant digestive tumors receiving active chemotherapy
  Interventions: Other: Food preference
- Patients with digestive cancer traited by immunotherapy: Patients with malignant digestive tumors receiving immunotherapy only
  Interventions: Other: Food preference

INTERVENTIONS:
Other: Food preference — Evaluate the impact of chemotherapy on the dietary preferences of patients with digestive cancer using a dietary and quality-of-life questionnaire at the beginning, middle and end of the chemotherapy/immunotherapy treatment.

SUMMARY:
Nutritional status is a major issue in the management of cancer patients. Forty to 60% of patients are undernourished at diagnosis. This undernutrition has a direct impact on patients' health and quality of life, with a reduction in survival associated with an increase in the risk of toxicity from anti-cancer treatments (chemotherapy, radiotherapy, surgery), the risk of infection and the risk of hospitalization. Thus, it is estimated that 10-20% of cancer patients die from the consequences of their undernutrition rather than from the tumor itself (Muscaritoli et al. 2021).

It is therefore recommended to systematically implement a multimodal nutritional intervention in cancer patients (recommendations of the learned societies ESPEN, ESMO and ASCO), combining nutritional support (oral and/or enteral and/or parenteral) with physical exercise (Muscaritoli et al. 2021). However, despite the systematic provision of dietary management, the effectiveness of nutritional interventions varies from patient to patient in terms of nutritional status, quality of life and overall survival (Cintoni et al. 2023).

Among the factors impacting patient compliance with dietary measures and their efficacy, sensory alterations occurring under chemotherapy potentially have a major impact (Drareni et al., 2019).

Indeed, the vast majority of patients describe an alteration in tastes and smells after starting chemotherapy treatment. However, few studies have focused on the specific parameters associated with these alterations. The aim of this study is to prospectively assess changes in sensory perceptions and eating habits in patients undergoing chemotherapy for digestive cancer at the start of treatment and after the first cycle of chemotherapy, and to correlate these alterations with patients' nutritional profile and clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete the proposed questionnaires
* Patients over 18 years of age
* Non-opposed patients
* Digestive cancers starting chemotherapy and/or immunotherapy
* Able to eat by mouth

Exclusion Criteria:

* Concomitant treatment for a non-digestive cancer (excluding basal/spinocellular carcinoma and chronic haemopathy)
* Previous ENT surgery (face/neck)
* Exclusive enteral feeding (nasogastric tube, gastrostomy) or parenteral nutrition
* Previous chemotherapy/immunotherapy < 5 years
* Individuals deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant digestive tumors receiving active chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient with changes in food preferences of digestive cancer patients at the end of the first cycle of chemotherapy. | At two month (end of the first cycle of chemotherapy/immunotherapy)
  Proportion of patients with 'altered' food preferences at the end of the first cycle of chemotherapy, with alteration defined as a reported decrease in appreciation for at least 30% of foods compared to before chemotherapy initiation

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Lyon Sud, Oullins-Pierre Bénite, France
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Croix Rousse, Lyon

IPD SHARING:
Plan to Share IPD: No